CLINICAL TRIAL: NCT03944356
Title: BRAF-/MEK-Inhibition With Dabrafenib and Trametinib in Melanoma Patients in the Adjuvant Setting: a Non-interventional Observatory Study
Brief Title: BRAF-/MEK-Inhibition With Dabrafenib and Trametinib in Melanoma Patients
Acronym: Combi-EU
Status: Completed | Type: Observational
Sponsor: EuMelaReg gGmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: EUMR-18001
Record Dates: First submitted 2019-04-26; First posted 2019-05-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dabrafenib and Trametinib — Dabrafenib and trametinib treatment under routine conditions according to the applying SmPC.
  Other Names: Tafinlar and Mekinist

SUMMARY:
Adjuvant therapy with dabrafenib plus trametinib in melanoma was approved in 2018 by the EMA (EUropean Medicines Agency).

The purpose of this non-interventional study is to assess the usage of adjuvant dabrafenib and trametinib in clinical practice, where the patient population may differ from study population.

DETAILED DESCRIPTION:
Melanoma is a disease of significant metastatic potential if not detected very early. Oncogenic mutations in BRAF (B-Raf proto-oncogene, serine/threonine kinase) are found in approximately 40% of melanomas and result in constitutive activation of the MAPK (Mitogen-Activated Protein Kinase) pathway.

Treatment with the BRAF inhibitor dabrafenib plus the MEK (Mitogen-activated protein kinase kinase) inhibitor trametinib showed improved overall survival in patients with unresectable or metastatic BRAF V600E/K-mutant melanoma (COMBI-d and COMBI-v studies). In an adjuvant setting treatment with dabrafenib and trametinib significantly reduced the risk of melanoma recurrence in patients with high-risk, stage III BRAF V600-mutant melanoma, with improvements in OS (Overall Survival), DMFS (Distant Metastasis Free Survival), and FFR (Freedom From Relaps) (COMBI-AD study). Based on these results, adjuvant dabrafenib plus trametinib therapy was approved in 2018 by the EMA.

Compared to the metastatic situation, issues of compliance and treatment adherence may be more relevant in adjuvant treatments, as patients are free of disease and potentially cured even without adjuvant treatment. As the routine administration of drugs including dosing, treatment interruptions, and early termination in clinical practice may vary from procedures defined in clinical trials, this study aims to assess the usage of adjuvant dabrafenib and trametinib in the routine clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete surgical resection of histologically confirmed AJCC (American Joint Committee on Cancer) (8th edition) clinical stage III (IIIA, IIIB, IIIC, IIID) melanoma, for whom a decision for adjuvant treatment with dabrafenib and trametinib has been made before entering the study.
* V600E/K mutation-positive cutaneous melanoma
* Adjuvant treatment with combination therapy of Dabrafenib (Tafinlar®) and Trametinib (Mekinist®) as indicated in the SmPC (Summary of Product Characteristics) and by prescription, that has been started no longer that 4 weeks before inclusion of the patient into the study or which will be initiated directly after inclusion
* Age ≥ 18 years
* Signed written informed consent

Exclusion Criteria:

* Lack of basic demographics and staging information
* Current or planned participation within a clinical trial. The participation in a follow-up phase of a clinical trial without active intervention is allowed.
* Current or planned treatment of another tumor disease except keratoacanthoma, squamous cell or basal cell carcinoma of the skin

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with complete surgical resection of histologically confirmed AJCC (8th edition) clinical stage III (IIIA, IIIB, IIIC, IIID) BRAF V600-mutated cutaneous melanoma who are planned to be treated or who already started treatment no longer than 4 weeks prior to study inclusion with dabrafenib and trametinib under routine conditions according to the applying SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Median time on treatment | Date of first dose up to 12 months
  Median time on adjuvant dabrafenib + trametinib treatment defined as the interval between start of treatment and permanent discontinuation of treatment.

SECONDARY OUTCOMES:
Permanent study drug discontinuation due to any reason | From date of first treatment until the date of treatment end, assessed up to 12 months
  Rate of permanent study drug discontinuation due to any reason.
Permanent study drug discontinuation due to adverse drug reactions | From date of first treatment until the date of treatment end, assessed up to 12 months
  Rate of permanent study drug discontinuation due to adverse drug reactions (ADRs).
Pyrexia and related symptoms | From date of first treatment until the date of treatment end, assessed up to 12 months
  Occurrence of pyrexia and related symptoms, listing the grade, number of episodes, and time to resolution.
Adverse drug reaction management: pyrexia | From date of first treatment until the date of treatment end, assessed up to 12 months
  Type of adverse drug reaction (ADR) management applied for pyrexia and correlation with occurrence/persistence of pyrexia.
Adverse drug reactions in Follow-up | From date of first treatment until the date of treatment end plus 3 months of follow-up, assessed up to 15 months
  ADRs persisting/emerging up to 3 months post-treatment.
Health-related quality of life | Over the course of treatment plus 3 months safety follow up, assessed up to 15 months
  Assessment of health-related quality of life (HRQoL), measured by the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC-QLQ-C30).
  The EORTC QLQ-C30 consists of the folowing scales, with each dimension specifying five levels of severity [not at all (level 1), a little (level 2), quite a bit (level 3), very much (level 4)]:
  * functional scales (Physical, Role, Cognitive, Emotional, Social Functioning)
  * symptom scales (Fatigue, Pain and Nausea/Vomiting)
  * single item scales (Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhoea and Financial Difficulties).
  Additionally the Global Health Status and QoL scales are incorporated, specifying on a scale from 1 (very poor) to 7 (excellent).
Relapse free survival | From date of first treatment until the date of treatment end, assessed up to 12 months
  Relapse free survival (RFS) time and rate
Distant metastasis free survival time | From date of first treatment until the date of treatment end, assessed up to 12 months
  Distant metastasis free survival (DMFS) time.
Distant metastasis free survival rate | From date of first treatment until the date of treatment end, assessed up to 12 months
  Distant metastasis free survival (DMFS) rate.
Overall survival time | From date of first treatment until the date of treatment end, assessed up to 12 months
  Overall survival (OS) time.
Overall survival rate | From date of first treatment until the date of treatment end, assessed up to 12 months
  Overall survival (OS) rate.
Time on treatment and efficacy endpoints | From date of first treatment until the date of treatment end, assessed up to 12 months
  Correlation between time on treatment and efficacy endpoints (RFS, DMFS, OS).

CONTACTS AND LOCATIONS:
Locations (36):
- Germany (36):
  - Elbe Kliniken Stade - Buxtehude GmbH, Buxtehude, Lower Saxony
  - Universitätsklinikum Essen, Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Essen, North Rhine-Westphalia
  - Universitätsklinik Kiel, Klinik für Dermatologie, Venerologie und Allergologie, Kiel, Schleswig-Holstein
  - Katholisches Klinikum Bochum, Bochum
  - Klinikum Bremen Mitte gGmbH, Bremen
  - Klinikum Bremerhaven Reinkenheide gGmbH, Bremerhaven
  - DRK Krankenhaus Chemnitz Rabenstein, Chemnitz
  - Klinikum Darmstadt GmbH, Darmstadt
  - Klinikum Dortmund gGmbH, Dortmund
  - Krankenhaus Dresden-Friedrichstadt, Dresden
  - Universitätsklinik Dresden, Dresden
  - HELIOS St. Johannes Klinik Duisburg, Duisburg
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitätsklinikum Greifswald, Greifswald
  - Universitätsklinik Halle, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Ludwigshafen gGmbH, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinik Magdeburg, Magdeburg
  - Universitaetsklinikum Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der Universität München, München
  - Fachklinik Hornheide, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Universitätsklinikum Regensburg, Regensburg
  - HELIOS Kliniken Schwerin, Schwerin
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm